CLINICAL TRIAL: NCT03293693
Title: Beta-glucan and Blood Glucose
Brief Title: Intake of Beta-glucan and Postprandial Regulation of Blood Glucose Metabolism in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Mills DA (Industry); Nofima (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016/648
Record Dates: First submitted 2017-03-10; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Post Prandial Blood Glucose; Gut Microbiota; Satiety
Keywords: beta-glucan; Blood glucose; Gut microbiota; Satiety; Dietary intervention
MeSH Terms: interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: Intervention With cross-over design. Three test meals will be tested.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test meal 1 (Experimental): Test meal with 0.5 g beta-glucan
  Interventions: Other: 0.5 g beta-glucan
- Test meal 2 (Experimental): Test meal with 3.5 g beta-glucan
  Interventions: Other: 3.5 g beta-glucan
- Test meal 3 (Experimental): Test meal with 8 g beta-glucan
  Interventions: Other: 8 g beta-glucan

INTERVENTIONS:
Other: 0.5 g beta-glucan — Dietary cross-over study with beta-glucan fiber
  Arms: Test meal 1
Other: 3.5 g beta-glucan — Dietary cross-over study with beta-glucan fiber
  Arms: Test meal 2
Other: 8 g beta-glucan — Dietary cross-over study with beta-glucan fiber
  Arms: Test meal 3

SUMMARY:
The overall aim is to investigate the intake of beta-glucan in relation to glucose metabolism and satiety in a postprandial study with healthy subjects. The potential effects will be related to changes in the gut microbiota, the circulating levels of short chain fatty acids, inflammation and gene expression in peripheral mononuclear blood cells

DETAILED DESCRIPTION:
The intervention study will have a fixed order, cross-over design with three test meals containing low (0.5 g / 100 g of product), medium (3.5 g / 100 g of product) and high (8 g / 100 g product) amount of beta -glucans, respectively. The test meals are in the form of cereals. All participants will eat the three test meals three constitutive days with 2 weeks apart. At day four, the participants will perform a postprandial glucose test (OGTT, 75 g glucose in 150 ml water) at Oslo and Akershus University College. Blood samples will be taken before and at different time points after glucose test.

At the screening visit the participants will be asked to limit the intake of dietary fiber from grains two weeks prior to the baseline visit (0) and during the study. Otherwise, participants will be asked not to change their diet and exercise habits during the study period.

At the baseline visit (visit 0) an OGTT will be performed. OGTT will also be performed at visit 1, 3 and 5 after intake of low, medium and high beta-glucan, respectively.

The participants will receive the test meals at visit 1, 2 and 4.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18,5 and 27 kg/m2
* Fasting plasma glucose ≤ 6.1 mmol/l

Exclusion Criteria:

* Chronic metabolic diseases such as diabetes type 1 and 2, coronary heart disease and cancer the last 6 months.
* Intestinal diseases such as chrons disease, ulcerative colitis and irritable bowel syndrome.
* Food allergy and intolerances towards grain and dairy products.
* Pregnant and lactating
* Smokers
* Fasting blood glucose ≥ 6.1 mmol/L
* CRP > 10 mg/L, measured at baseline (visit 0)
* BMI <18,5 and >27 kg/m2
* Planned weight reduction and or ± 5% weight change over the past three months.
* Use of antibiotics last 3 months before study entry and during the study period
* Use of probiotics the last month before study entry and during the study period
* Blood donor last 2 months before study entry and or during the study period
* Not willing to end the use of dietary supplements four weeks prior to study entry and throughout the study period
* Alcohol consumption > 40g / day
* Hormone treatments (except contraceptives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose response | At day 4
  Blood glucose response after OGTT
Postprandial insulin response | At day 4
  insulin response after OGTT

SECONDARY OUTCOMES:
H2 breath response | At day 4
  H2 breath response after OGTT
Free fatty acids | At day 4
  Plasma free fatty acids are measured after intake of test meals
Microbiota analyses in feces | At day 4
  Microbiota analyses in feces are measured before and after intake of test meals. Change in microbiota will be analysed
Serum triglyceride response | At day 4
  Triglyceride response are measured are measured after OGTT
Serum cholesterol | At day 4
  Serum cholesterol are measured fasting after intake of test meals
hunger and satiety hormones (e.g. GLP1) | At day 4
  The response in hunger and satiety hormones after OGTT
Inflammatory markers (e.g. CRP) | At day 4
  Response in Inflammatory markers are measured after OGTT
mRNA analyses in PBMC (RT-PCR) | At day 4
  PBMC are collected before and after OGTT. The change in mRNA level will be analyzed
Quantitative assessment of metabolites in urine | At day 4
  Morning urine are collected before and after intake of test meals. Metabolites in urine will be quantified using UHPLC-qTOF-MS. Change in metabolites before and after test meals will be analyzed
Quantitative assessment of metabolites in plasma | At day 4
  Plasma for metabolome analyses are collected after intake of test meals. Metabolites in plasma will be quantified using UHPLC-qTOF-MS.
Visual analogue scale (VAS) | At day 1
  Subjective hunger and satiety will be estimated after intake of test meals for one day
Visual analogue scale (VAS) | At day 3
  Subjective hunger and satiety will be estimated after intake of test meals for three days

CONTACTS AND LOCATIONS:
Overall Officials: Mari CW Myhrstad, PhD, Principal Investigator — Oslo and Akershus University College
Locations (1):
- Oslo and Akershus university College, Oslo, Norway

REFERENCES:
- [Derived] Telle-Hansen VH, Gaundal L, Hogvard B, Ulven SM, Holven KB, Byfuglien MG, Mage I, Knutsen SH, Ballance S, Rieder A, Rud I, Myhrstad MCW. A Three-Day Intervention With Granola Containing Cereal Beta-Glucan Improves Glycemic Response and Changes the Gut Microbiota in Healthy Individuals: A Crossover Study. Front Nutr. 2022 Apr 28;9:796362. doi: 10.3389/fnut.2022.796362. eCollection 2022. PMID 35578615